CLINICAL TRIAL: NCT05533229
Title: Fentanyl Versus Morphine in Spinal Anesthesia for Caesarian Section - Study on Perioperative Analgesia, Side Effects and Patient 's Satisfaction
Brief Title: Fentanyl Versus Morphine in Spinal Anesthesia for Caesarian Section - Study on Analgesia, Side Effects and Patient 's Satisfaction
Acronym: FvMinSA
Status: Completed | Type: Observational
Sponsor: Dr. Mihai Octavian Botea (Other)
Collaborators: Oradea Pelican Clinic Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Mihai Octavian Botea, MD, PhD, Assistant professor, University of Oradea
Organization: University of Oradea (Other)
Other Study IDs: 07FvM_Medical Study
Record Dates: First submitted 2022-07-10; First posted 2022-09-08 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia
Keywords: spinal anesthesia, pain scores, spinal opioids side effects, patient's satisfaction
MeSH Terms: interventions — Fentanyl; Bupivacaine; Morphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant patients scheduled for C section: Spinal anesthesia
  Interventions: Drug: Fentanyl; Drug: Morphine

INTERVENTIONS:
Drug: Fentanyl — The trial aims to study the quality of anesthesia and perioperative analgesia and patient's satisfaction provided by fentanyl and bupivacaine versus morphine and bupivacaine.
  Other Names: plus Bupivacaine
Drug: Morphine — The trial aims to study the quality of anesthesia, perioperative analgesia and patient's satisfaction provided by fentanyl and bupivacaine versus morphine and bupivacaine.
  Other Names: plus Bupivacaine

SUMMARY:
Intrathecal morphine and fentanyl are used for anesthesia and perioperative pain management in caesarian section. Despite the fact that spinal Fentanyl is better tolerated, might not be enough for postoperative pain control. Morphine offers an improved analgesia but might be not tolerated due to a higher incidence of side effects, especially nausea and vomiting.

This is a prospective, randomized, double-blind, parallel study including 80 parturients scheduled for elective CS. Spinal anesthesia is consisting in bupivacaine (7.5 - 10 mg in relation to height) and either fentanyl 25 mcg (F group) either morphine 100 mcg (m group). It will be assessed intraoperative and postoperative pain scores, the incidence of sides effects, patient's satisfaction and systemic opioids consumption.

DETAILED DESCRIPTION:
The patients were randomly allocated into one of the two groups M (morphine) or F (fentanyl) with a sample size calculation at 1:1 ratio, using the envelope technique.

Group F (fentanyl) was administered hyperbaric bupivacaine 0.5% along with a standard dose of 25 mcg fentanyl, while group M (morphine) received hyperbaric bupivacaine 0.5% with a standard dose of 100 mcg morphine. The dose of hyperbaric bupivacaine 0.5% to be injected, was based on the patient's height and here were used a range of doses between 7.5 mg and 11 mg.

The study required two anesthetists. The first anesthetist was "in charge" and performed the spinal anesthesia and he was blind to the solution used. The second anesthetist randomly assigned the patient, drew up the intrathecal solution and provided the anesthetic mixture. By this method, the first anesthetist was totally blinded to the opioid used. All drugs were from the same manufacturer.

During the pre-anesthetic visit, the patient received information about the aims of the study, the method of anesthesia, and details about the pain management and about the pain assessment with the numeric pain scale (NPS). Patient's demographics data were obtained: height, term weight and age. Also, full medical past and drugs history, previous allergies and other important medical data were documented.

Pre-operatively a venous access was obtained with an 18 G. cannula and 500 ml of Ringer lactate solution was infused prior to anesthesia. Participants were fasting and received pantoprazol 40 mg and metoclopramide 10 mg as pre-anesthetic medication. The spinal anesthesia was performed in an aseptic technique with the patient in a sitting position, in the L3 - L4 interspace, using a midline approach, with a Whitacre 27 G. needle and the anesthetic mixture manually injected at a rate of 1 ml.15s-1, with a barbotage effect. A previous skin local anesthetic infiltration was performed with 2 ml of 1% lidocaine. After the block, the patient was placed in a supine position with a roll wedge placed under the right hip to displace the uterus to the left until fetal extraction. Volemic supply was assured with warm Ringer lactate (10-20 ml.kg-1hr-1). All patients than had anti-embolic socks on lower limbs.

Surgery started when sensory block, as assessed by the cold test, reached the T4 dermatome level.

Non-invasive blood pressure (BP) was measured every minute until the baby was delivered and every 3-5 minutes afterwards. Any decrease in systolic blood pressure below the background level resulted in intravenous ephedrine and doses of 5-15 mg being given, repeated every minute until the systolic blood pressure had been restored. At delivery, oxytocin 5 I.U. was given intravenously (normal practice when the study was conducted) and afterwards as required.

We took a proactive action to prevent the perianesthetic emetic syndrome. So, our patients received from the time of surgery a nausea prophylaxis with granisetron 1 mg and a dose o dexamethasone 4 mg. A second dose of granisetron 1 mg was given at 12 hours apart. Afterwards only as required anti-emetic medication was given.

Heart rate, BP, oxygen saturation as measured by pulse oximetry (SpO2), requirement for supplemental analgesics, need for conversion to general anesthesia were recorded intraoperatively. In addition to these parameters, the level of sensory block was assessed by the cold test, and the maximum motor block score was recorded using a 4-points Bromage scale as the complete motor recovery time.

The postoperative pain control strategy was relaying on regular paracetamol 1 gr., every 6 hrs. and ibuprophen 400 mg every 8 hrs., both drugs given in intravenous or oral administration. As required for breakthrough pain, were available doses of 50 to 100 mg. of iv. tramadol, 6 hourly to a maximum dose of 400 mg.

Data collection We collected data regarding: demographics (age, weight, height, smoke consumption, gesta/para status and preoperative contractions); time from anesthesia to incision; time to sensory block; pain scores (at surgical incision, end of surgery, at 4 h, 6 h, 12 h, 24 h, 48 h, 72 h - postoperative the pain scores were assessed at rest and on mobilizing); AUE72h (sum pain intensity differences area over 72 hours) and SPID72h (time-weighted sum pain intensity differences over 72 hours); side effects associated with anesthesia (pruritus with a grading scale, nausea, vomiting, over sedation, dizziness and respiratory depression).

Contribution to pain intensity assessment metrics Besides assessing and understanding the level of pain, pain scales help healthcare practitioners to make a well-informed and accurate diagnoses as well as to formulate carefully-considered treatment plan for their patients.

The Numeric Pain Rating Scale is a type of unidimensional pain scale which comes with numbers, from 0 to 10. A person simply needs to rate their pain based on written or verbal prompts, from 0 meaning no pain to 10 meaning worst pain imaginable.

But for a more comprehensively comparison of the post-operative pain in the study groups, two additional assessment metrics were employed:

1. time-weighted sum pain intensity differences over 72 hours
2. sum pain intensity differences area over 72 hours Descriptive statistics included the observed frequency counts (percentage) for categorical variables; and mean ± standard deviation for numerical variables, irrespective of their distribution. Normality was tested with the Kolmogorov-Smirnov test. For comparing means in normally distributed values, the t-test for independent samples was applied, with Levene's test for equality of variances. For comparing distribution of non-normally distributed numerical values, the non-parametric Mann-Whitney U statistical tests was applied and median (Inter-Quartile Range) with Tukey's hinges was additionally provided as a descriptive statistic.

The Chi-square statistical test (either asymptotic, Fisher's exact test, or Monte-Carlo simulation with 10,000 samples) was applied to check the statistical significance of the association between the categorical variables. The odds ratio (OR) values were calculated for the symptoms associated with the two anesthetics, such as nausea and dizziness.

The statistical analysis was conducted at a 95% level of confidence and a 5% level of statistical significance. All reported probability values were two-tailed.

Statistical analysis was performed with the statistical software IBM SPSS v. 20 and open source R v.4.0.5 packages.

Ethics The study was conducted in accordance with the Declaration of Helsinki, and the protocol was approved by the Ethics Committees of Pelican Hospital from Oradea (no.2672/28.12.2021).

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* no medical past history
* not known allergies to the used medication
* no history of chronic pain ar regular use of analgesics
* no past history of anxiety or depression
* body weight ≥ 50 kg
* elective C section indication
* single fetus

Exclusion Criteria:

* conversion from a natural delivery with/without an epidural anesthesia started
* pregnant women with psychiatric disorder;
* history of drug addiction; diagnosis of acute or chronic fetal distress; contraindication of spinal anesthesia;
* patient refusal;
* preeclamptic patients, patients who developed allergic reaction after enrolling in the study;
* refusal of the pain killers or other protocol medication prescribed;
* the necessity of surgical reintervention in the next 72 h after C-section;
* previous administration of opioids and/or other central nervous system depressants.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — study's population is the pregnant woman
Study Population: The study population will be selected from the pregnant patients of Oradea Pelican Clinic Hospital.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
to assess the perioperative analgesia using Numeric Pain Scale | 6 months
  assessing pain scores (at surgical incision, end of surgery, at 4 h, 6 h, 12 h, 24 h, 48 h, 72 h - postoperative the pain scores were assessed at rest and on mobilization); AUE72h (sum pain intensity differences area over 72 hours) and SPID72h (time-weighted sum pain intensity differences over 72 hours); the pain scores according to the Numeric Pain Scale it will be rated between 0 and 10, meaning 0 - no pain and 10 - the worst pain imaginable
assessing the degree of patient's of satisfaction | 6 months
  assessing the degree of satisfaction on a five point scale with the highest rate as being "completely satisfied", followed by "satisfied", "so so", "unsatisfied" and "completely usatisfied"

SECONDARY OUTCOMES:
to assess the incidence of and degree of pruritus as a side effect related to intrathecal opioids | 6 months
  it will be assessed the presence of pruritus and it's degree on a 4 point scale as follows: 0 - absent, 1 - minor, 2 - moderate, 3 - severe.
to assess the incidence of other side effects related to intrathecal opioids | 6 months
  to assess the incidence of other side effects like: nausea, vomiting, dizziness, sedation and respiratory depression; regarding this secondary outcome measure it will be assessed as present or not during the 72 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Bimbo-Szuhai, MD PhD, Study Chair — Head of Anesthesia Department at Oradea Pelican Clinic Hospital
Locations (1):
- University of Oradea, Pelican Clinic Hospital, Oradea, Bihor County, Romania

REFERENCES:
- [Result] Fonseca NM, Guimaraes GMN, Pontes JPJ, Azi LMTA, de Avila Oliveira R. Safety and effectiveness of adding fentanyl or sufentanil to spinal anesthesia: systematic review and meta-analysis of randomized controlled trials. Braz J Anesthesiol. 2023 Mar-Apr;73(2):198-216. doi: 10.1016/j.bjane.2021.10.010. Epub 2021 Dec 24. PMID 34954261
- [Result] Karaman S, Gunusen I, Uyar M, Biricik E, Firat V. The effects of morphine and fentanyl alone or in combination added to intrathecal bupivacaine in spinal anesthesia for cesarean section. Agri. 2011 Apr;23(2):57-63. PMID 21644105
- [Result] Weigl W, Bierylo A, Wielgus M, Krzemien-Wiczynska S, Kolacz M, Dabrowski MJ. Perioperative analgesia after intrathecal fentanyl and morphine or morphine alone for cesarean section: A randomized controlled study. Medicine (Baltimore). 2017 Dec;96(48):e8892. doi: 10.1097/MD.0000000000008892. PMID 29310376
- [Result] Seki H, Shiga T, Mihara T, Hoshijima H, Hosokawa Y, Hyuga S, Fujita T, Koshika K, Okada R, Kurose H, Ideno S, Ouchi T. Effects of intrathecal opioids on cesarean section: a systematic review and Bayesian network meta-analysis of randomized controlled trials. J Anesth. 2021 Dec;35(6):911-927. doi: 10.1007/s00540-021-02980-2. Epub 2021 Aug 2. PMID 34338864
- [Result] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Result] Overall JE, Shobaki G, Shivakumar C, Steele J. Adjusting sample size for anticipated dropouts in clinical trials. Psychopharmacol Bull. 1998;34(1):25-33. PMID 9564195
- [Result] Stewart WC, Jackson AL, Jenkins JN. Dropout rates for intent-to-treat and per protocol analyses. Am J Ophthalmol. 2004 Apr;137(4):639-45. doi: 10.1016/j.ajo.2003.11.028. PMID 15059702
- [Result] Girgin NK, Gurbet A, Turker G, Aksu H, Gulhan N. Intrathecal morphine in anesthesia for cesarean delivery: dose-response relationship for combinations of low-dose intrathecal morphine and spinal bupivacaine. J Clin Anesth. 2008 May;20(3):180-5. doi: 10.1016/j.jclinane.2007.07.010. PMID 18502360
- [Result] Mallick-Searle T, Fillman M. The pathophysiology, incidence, impact, and treatment of opioid-induced nausea and vomiting. J Am Assoc Nurse Pract. 2017 Nov;29(11):704-710. doi: 10.1002/2327-6924.12532. PMID 29131554